CLINICAL TRIAL: NCT03905447
Title: An Open-label, Pilot Study to Assess Safety, Tolerability, Pharmacokinetics and Effects of Inhaled PC945 in the Pre-emptive Treatment of Aspergillus Fumigatus Colonisation in Lung Transplant Recipients
Brief Title: The Effect of Early Treatment of PC945 on Aspergillus Fumigatus Lung Infection in Lung Transplant Patients.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study is being terminated early as a result of the coronavirus (COVID-19) outbreak.
Sponsor: Pulmocide Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PC_ASP_002; 2018-000240-26 (EudraCT Number)
Record Dates: First submitted 2019-03-06; First posted 2019-04-05 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2020-06

CONDITIONS: Aspergillosis; Lung Transplant Infection
MeSH Terms: conditions — Aspergillosis | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Subjects in the surveillance phase with detectable Aspergillus fumigatus lung infections WITHOUT clinical symptoms will be eligible to receive PC945 for 28 days. Following 28 days on PC945, subjects with ongoing A. fumigatus lung infections may receive a further 56 days of PC945.
  Subjects in the surveillance phase with EITHER detectable Aspergillus fumigatus lung infections WITH clinical symptoms, OR other fungal lung infection, will be eligible to be followed up for 16 weeks on Standard of Care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PC945 (Experimental)
  Interventions: Drug: PC945
- Standard of Care (Other): Standard of care anti-fungal medication
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: PC945 — Nebulized PC945 5mg OD for 28 days with an optional extended treatment period of a further 56 days.
  Arms: PC945
Drug: Standard of Care — Standard of Care antifungal medication
  Arms: Standard of Care

SUMMARY:
This study tests the effects of pre-emptive treatment with an experimental drug PC945 in lung transplant recipients whose lungs are infected by the fungus Aspergillus fumigatus.

PC945 may be useful in treating patients infected with Aspergillus fumigatus as, unlike the usual treatments, it is inhaled into the lung and has been designed to stay there and treat the infection. Participants will be monitored for up-to 12 weeks for the presence of Aspergillus in their lungs. Suitable participants will receive PC945 for an initial 28 days (Pre-emptive treatment phase) and, if needed, a further 8-weeks (Extended treatment phase).The amount of fungus in the patients' lungs will be measured over the course of the study. Participants with lung infections but not eligible for PC945 will be followed-up for 16-weeks on standard of care treatment. The study will take place at multiple sites in UK and 10 participants will receive PC945. The maximum study duration will be about 28 weeks.

ELIGIBILITY:
Inclusion Criteria (Surveillance Phase)

* Between the ages of 18 and 85 years.
* Received a single or bilateral lung transplant.
* Provided written informed consent prior to transplant

Exclusion Criteria (Surveillance Phase)

* Is precluded from participating in this study as a result of treatment with another investigational drug or participation in another clinical trial.
* If female, the subject is pregnant, lactating or breast feeding.
* Any other clinically significant disease or condition, which in the Investigator's medical opinion would preclude the subject's participation in a clinical trial (e.g., recent myocardial infarction).
* Is employed or is a first-degree relative of anyone employed by Pulmocide, a participating clinical trial site, or any contract research organisation involved in the study.
* Is receiving antiretroviral protease inhibitor therapy.
* Has human immunodeficiency virus or chronic, active hepatitis infection, or had a positive hepatitis B surface antigen or hepatitis C virus RNA test prior to transplant.
* Any known history or current evidence of alcohol or drug abuse that, in the Investigator's opinion, would exclude the subject from participation in the study

Inclusion Criteria (Pre-emptive Treatment Phase)

* A positive test for A. fumigatus in BAL during the Surveillance Phase of the study
* Provided written informed consent for participating in the Pre-Emptive Treatment Phase.

Exclusion Criteria (Pre-emptive Treatment Phase)

* Clinical, endobronchial and/or radiological features of fungal disease.*
* Any other disease or condition, which in the Investigator's medical opinion would preclude the subject's participation in the Pre-Emptive Treatment Phase of the study (e.g., recent myocardial infarction).

Inclusion Criteria (Follow-up Phase - SOC Antifungal Treatment)

* Subject is not eligible to receive pre-emptive PC945 treatment due to either clinical, endobronchial and/or radiological features of fungal disease OR a fungal infection other than A. fumigatus in BAL, that requires SoC antifungal treatment to be started during the Surveillance Phase of the study.
* Provided written informed consent for participating in the Follow-Up Phase for SoC antifungal treatment.

Exclusion Criteria (Follow-up Phase - SOC Antifungal Treatment)

* Any other disease or condition, which in the Investigator's medical opinion would preclude the subject's participation in the Follow-Up Phase for SoC antifungal treatment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) | 48 hours Post Transplant to Week 16 post treatment
Proportion of participants receiving PC945 who meet the markedly abnormal criteria for 12-lead ECG assessment at lease once post dose | Baseline to Week 16
Proportion of participants receiving PC945 who meet the markedly abnormal criteria for vital signs assessment at lease once post dose | Baseline to Week 16
Proportion of participants receiving PC945 who meet the markedly abnormal criteria for safety laboratory assessment at lease once post dose | Baseline to Week 16
Predicted post bronchodilator forced expiratory volume in 1 second (FEV1) values from participants receiving PC945 | Baseline to Week 16
Forced vital capacity (FVC) values from participants receiving PC945 | Baseline to Week 16
Area under the curve from time 0 to 2 h post-dose (AUC0-2) | Baseline to Week 16
  Derived pharmacokinetic parameters for PC945 and the potential circulating metabolite(s), if detectable
Maximum plasma concentration | Baseline to Week 16
  Derived pharmacokinetic parameters for PC945 and the potential circulating metabolite(s), if detectable
Concentration at the end of the dosage interval (Ctrough) | Baseline to Week 16
  Derived pharmacokinetic parameters for PC945 and the potential circulating metabolite(s), if detectable

SECONDARY OUTCOMES:
Lung Concentration of PC945 | Baseline to Week 16
A. fumigatus fungal culture status (presence or absence) in subjects with a baseline A. fumigatus-positive bronchoalveolar lavage (BAL) | Baseline to Week 16
Change in BAL A. fumigatus measured by quantitative polymerase chain reaction (qPCR) | Baseline to Week 16
Change in the number of sputum A. fumigatus colony forming units (CFU) in cultured BAL. | Baseline to Week 16
Galactomannan levels in BAL | Baseline to Week 16
Aspergillus status (Presence or absence) of BAL using an Aspergillus immunochromatographic lateral flow device (AspLFD). | Baseline to Week 16
Status of fungal hyphae or pseudohyphae (presence or absence) on cytological examination | Baseline to Week 16
Subject experience of inhaled PC945 | Baseline to Week 16
  Assessed by a standardised study-specific questionnaire assessing participants' subjective experience across a number of domains including taste, smell and overall acceptability following inhalation of PC945.
Subject experience of inhaled amphotericin B | Baseline to Week 16
  Assessed by a standardised study-specific questionnaire assessing participants' subjective experience across a number of domains including taste, smell and overall acceptability, following inhalation of amphotericin B.

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Papworth Hospital, Papworth Everard, Cambridge
  - Harefield Hospital, Harefield, Uxbridge
  - Wythenshawe Hospital, Manchester